CLINICAL TRIAL: NCT02920944
Title: Technical Feasibility and Diagnostic Yield of New 20-gauge Procore Needle for EUS-guided FNA Biopsy in Solid Pancreatic Lesions; Comparison With 22-gauge Procore Needle
Brief Title: Diagnostic Yield of 20-gauge Procore Needle for EUS-guided FNA Biopsy in Solid Pancreatic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seung Bae Yoon (Other)
Collaborators: Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Seung Bae Yoon, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EUS 20 gauge
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-FNB with 20-gauge (Experimental): EUS-FNB with 20-gauge procore needle
  Interventions: Device: EUS-FNB with 20 gauge ProCore needle
- EUS-FNB with 22-gauge (Active Comparator): EUS-FNB with 22-gauge procore needle
  Interventions: Device: EUS-FNB with 22 gauge ProCore needle

INTERVENTIONS:
Device: EUS-FNB with 20 gauge ProCore needle — EUS-FNB with 20-gauge (Echotip ProCore; Cook Endoscopy Inc, Limerick, Ireland)
  Arms: EUS-FNB with 20-gauge
Device: EUS-FNB with 22 gauge ProCore needle — EUS-FNB with 22-gauge (Echotip ProCore; Cook Endoscopy Inc, Limerick, Ireland)
  Arms: EUS-FNB with 22-gauge

SUMMARY:
This study aims to examine technical feasibility and diagnostic yield of new 20-gauge Procore needle for EUS-guided fine needle biopsy in solid lesions by comparing with 22-gauge Procore needle. The study design is prospective, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years referred to our medical center for EUS-FNB with diagnosed or suspected solid pancreatic masses according to clinical evaluation and imaging studies.

Exclusion Criteria:

* cystic pancreatic lesions, patients haemodynamically unstable or with severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 50,000 cells/cubic millimeter [cmm3]), patients unable to suspend anticoagulant/anti-platelet therapy, pregnancy, inability or refusal to give informed consent, and refusal to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
single diagnostic yield of the histologic core | up to 5 minutes after endoscopic ultrasound-guided fine needle biopsy

SECONDARY OUTCOMES:
total diagnostic yield of the histologic core | up to 5 minutes after endoscopic ultrasound-guided fine needle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: In Seok Lee, MD, Study Director — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul, No State, South Korea

IPD SHARING:
Plan to Share IPD: Undecided